CLINICAL TRIAL: NCT00075374
Title: A Multicenter, Randomized Phase II Study of Two Schedules of Taxotere (Weekly Versus Every 3 Weeks) in Elderly or Poor Performance (ECOG PS 2), Chemotherapy-Naive Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Two Regimens of Docetaxel in Treating Patients Who Have Not Received Chemotherapy For Unresectable Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSMC1503; CWRU-MSMC-1503; AVENTIS-GIA-12143; THERADEX-GIA-12143; MTSMC-LUN06
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel (Experimental)
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel — Patients receive docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  OR Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline, every 2 courses during study treatment, and then at study completion.
  Patients are followed at 1 month and then every 2-3 months thereafter.
  Other Names: Taxotere; Docefrez

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which docetaxel regimen is more effective for non-small cell lung cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of two regimens of docetaxel in treating patients who have not previously received chemotherapy for unresectable stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effects of two different schedules of docetaxel on the incidence of grade 3 and 4 toxic effects in older or poor performance chemotherapy-naïve patients with unresectable stage IIIB or IV non-small cell lung cancer.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the response rate in patients treated with these regimens.
* Compare the incidence of serious adverse events in patients treated with these regimens.
* Determine the quality of life of patients treated with these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 2 courses during study treatment, and then at study completion.

Patients are followed at 1 month and then every 2-3 months thereafter.

PROJECTED ACCRUAL: A total of 210-230 patients (105-115 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Unresectable stage IIIB or IV disease
* No untreated brain or leptomeningeal metastases

  * Treated patients must be neurologically stable and the adverse effects from prior therapy must be resolved to grade 2 or less after the completion of treatment
* No symptomatic (i.e., requiring thoracentesis) pleural effusion
* No clinically significant (i.e., grade 3 or greater) pericardial effusion

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 (70 years of age and over) OR
* ECOG 2 (under 70 years of age)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8.0 g/dL

Hepatic

* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal (ULN) if alkaline phosphatase is no greater than ULN OR
* Alkaline phosphatase no greater than 4 times ULN if ALT and AST are no greater than ULN

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No grade 2 or greater peripheral neuropathy
* No prior hypersensitivity reaction to taxanes or products containing polysorbate 80
* No other active malignancy except carcinoma in situ of the cervix or basal cell skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study treatment or follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Recovered from prior radiotherapy (i.e., side effects resolved to grade 2 or less)
* No concurrent radiotherapy

Surgery

* More than 3 weeks since prior major surgery

Other

* More than 30 days since prior anticancer investigational drugs

  * Concurrent supportive care investigational agents allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States